CLINICAL TRIAL: NCT01944098
Title: Systemic Intraoperative Lidocaine Infusion for Postoperative Pain Management in Obese Patients: A Randomized, Placebo-Controlled Pilot Study
Brief Title: Intraoperative Lidocaine Infusion for Postoperative Pain Management in Obese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00002417
Record Dates: First submitted 2013-08-12; First posted 2013-09-17 (Estimated); Results first posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2015-12

CONDITIONS: Bariatric Surgical Pain
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Experimental): Intraoperative continuous IV infusion of Lidocaine at 2mg/kg/hr
  Interventions: Drug: Lidocaine
- Placebo (Active Comparator): Intraoperative continuous placebo infusion of dextrose at 2mg/kg/hr
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine
  Arms: Lidocaine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to assess the feasibility and safety of administering continuous intraoperative lidocaine infusions in adult patients undergoing laparoscopic Roux en Y Gastric Bypass (RYGB). The secondary objective is to determine if lidocaine administration versus placebo (dextrose administration) (initiated at the time of anesthesia induction and continued until extubation) will reduce postoperative narcotic requirements.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 18-65 years old
* BMI ≥ 40 kg/m2, ≤ 60 kg/m2
* Undergoing a primary laparoscopic RYGB by Dr. Murr
* Agree to be followed 24 hours postoperatively
* Normal K+ and Mg++ serum levels

Exclusion Criteria:

* BMI less than 40 kg/m2, > 60 kg/m2
* Laparoscopic RYGB surgery performed by a surgeon other than Dr. Murr
* Allergy to lidocaine
* Allergy to hydromorphone or ketorolac
* Allergy to corn or amide anesthetics
* Use of (thioridizine)
* Pregnancy
* Abnormalities of ALT or AST
* Intra-operative diagnosis of cirrhosis or portal hypertension
* Intraoperative complications per surgeon
* Intraoperative extensive adhesions per surgeon
* Chronic pain syndrome and chronic use of narcotics
* Severe back pain secondary to degenerative joint disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Karlnoski, PhD, Study Director — Florida Gulf-to-Bay Anesthesiology
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine: Intraoperative continuous IV infusion of Lidocaine at 2mg/kg/hr
  Lidocaine
- Placebo: Intraoperative continuous placebo infusion of dextrose at 2mg/kg/hr
  Placebo
Period: Overall Study
Arm/Group | Lidocaine | Placebo
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Patients received 2mg/kg/hr of lidocaine intraoperatively from the time of induction until the time of emergence.
- Placebo Arm: Patients received 2mg/kg/hr of placebo (saline) intraoperatively from the time of induction until the time of emergence.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 47.3 (8.3) | 47.5 (7.4) | 47.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
BMI [Mean (Standard Deviation); unit: kg/m^2] | 46.4 (6.1) | 48.3 (5.6) | 47.5 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Analysis of patient outcome will involve a series of visual analogue scale pain evaluations during mobilization, coughing, and resting. VAS, 0 cm as no pain - 10 cm as maximum pain
Time Frame: 6 hours post-surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 9 | 10
units on a scale
  Resting VAS | 3 [0 to 10] | 4.5 [0 to 8]
  Coughing VAS | 8 [3 to 10] | 8 [5 to 9]
  Moving VAS | 8 [0 to 10] | 8 [4 to 9]

2. Primary Outcome: Postoperative Pain
Description: Analysis of patient outcome will involve a series of visual analogue scale (VAS, 0 cm as no pain - 10 cm as maximum pain) pain evaluations during mobilization, coughing, and resting
Time Frame: 12 hours post-surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 9 | 10
units on a scale
  Resting VAS | 3.5 [0 to 9] | 4 [0 to 6]
  Coughing VAS | 7 [5 to 10] | 7 [2 to 9]
  Moving VAS | 8 [5 to 10] | 7 [5 to 8]

3. Primary Outcome: Postoperative Pain
Description: as for outcome 2
Time Frame: 18 hours post-surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 9 | 10
units on a scale
  Resting VAS | 2.5 [0 to 9] | 4.5 [0 to 8]
  Coughing VAS | 6 [2 to 10] | 6.5 [4 to 9]
  Moving VAS | 6 [4 to 9] | 7 [4 to 8]

4. Primary Outcome: Postoperative Pain
Description: as for outcome 1
Time Frame: 24 hours post-surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 9 | 10
units on a scale
  Resting VAS | 3 [0 to 8] | 3.5 [0 to 10]
  Coughing VAS | 8 [2 to 10] | 5.5 [4 to 10]
  Moving VAS | 6 [2 to 10] | 4.5 [4 to 10]

ADVERSE EVENTS:
Time Frame: Within 1 hour post-operation
Description: The primary outcome was the presence of lidocaine toxicity symptoms at 1 hour after lidocaine infusion cessation. We defined this endpoint as numbness or a metallic taste in the tongue or mouth, dizziness, and/or lightheadedness as reported by the patient and objectively as blood pressure changes.
Arm/Group | Lidocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=10) | Placebo (N=10)
Dizziness (General disorders) | 1 (1) | 4 (4) — post-operation lightheadedness
Metallic Taste in Mouth (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Significant Blood Pressure Changes (Blood and lymphatic system disorders) | 0 (0) | 0 (0) — Postoperative blood pressure change that is greater than 20% from the baseline blood pressure measured preoperatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No